CLINICAL TRIAL: NCT00725764
Title: A Phase 2 Study of the MET RTK Inhibitor GSK1363089 (Formerly XL880) in Subjects With Recurrent or Metastatic Squamous Cell Cancer of the Head and Neck
Brief Title: Phase 2 Study of GSK1363089 (Formerly XL880) in Adults With Squamous Cell Cancer of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MET111646; NCT00482326 (obsolete NCT alias)
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-07

CONDITIONS: Neoplasms, Head and Neck
Keywords: VEGFR2; XL880; foretinib; Squamous Cell Cancer of the Head and Neck; MET; GSK1363089
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — GSK 1363089

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Participants who qualified for study entry received 240 mg of GSK1363089 (foretinib) on a 5-day on 9-day off schedule every 2 weeks.
  Interventions: Drug: GSK1363089 (foretinib)

INTERVENTIONS:
Drug: GSK1363089 (foretinib) — Multitargeted tyrosine kinase inhibitor
  Other Names: GSK1363089 (formerly XL880)

SUMMARY:
This study is being conducted to determine the best confirmed response rate, safety, and tolerability of GSK1363089 treatment in adult subjects with squamous cell carcinoma of the head and neck (SCCHN). GSK1363089 is a new chemical entity that inhibits multiple receptor tyrosine kinases (RTKs) with growth-promoting and angiogenic properties. The primary targets of GSK1363089 are the HGF and vascular endothelial growth factor (VEGF) RTK families (eg, MET, VEGFR2/kinase insert domain receptor [KDR]). Since MET overexpression has been associated with poorer prognosis and MET tyrosine kinase mutations have been reported in SCCHN, inhibition of MET receptor and VEGFR2/KDR activation by agents such as GSK1363089 may be of therapeutic benefit in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a histologically or cytologically confirmed diagnosis of SCCHN and
* has recurrent and/or metastatic disease
* is not eligible for curative intent surgery or radiotherapy
* has no history of uncontrolled tumor bleeding including hemoptysis in patients with documented pulmonary metastasis.
* The subject has measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as =20 mm with conventional techniques, or as =10 mm with spiral computerized tomography (CT) scan.
* Subject is capable of swallowing capsules.
* Fifteen unstained slides of tumor tissue, archival or fresh, or paraffin block are available, and there - confirmation that samples have been sent for analysis at the central laboratory.
* The subject is at least 18 years old.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status =1.
* In the adrenocorticotropic hormone (ACTH) stimulation test, the subject has a serum cortisol level =20 µg/dL (552 nmol/L) 30-90 minutes after injection of ACTH.
* The subject has organ and marrow function as follows: absolute neutrophil count (ANC) =1500/mm3, platelets =100,000/mm3, hemoglobin =9 g/dL, bilirubin =1.5 mg/dL, serum creatinine =1.5 mg/dL and/or calculated creatinine clearance =60 mL/min, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =2.5 times the upper limit of normal if no liver involvement or =5 times the upper limit of normal with liver involvement.
* The subject has signed the informed consent document.
* Sexually active subjects must use a medically accepted method of contraception during the course of the study.
* Female patients of childbearing potential must have a negative pregnancy test at enrollment.
* The subject has had no other diagnosis of malignancy (unless non-melanoma skin cancer, in situ carcinoma of the cervix, or a malignancy diagnosed =5 years ago, and has had no evidence of disease for 5 years prior to screening for this study).

Exclusion Criteria:

* The subject has received radiation to >25% of his or her bone marrow within 30 days of GSK1363089 treatment.
* The subject has received an investigational drug within 30 days (or <5.5 half lives) of the first dose of study drug.
* The subject has received more than one regimen of systemic anticancer therapy for disease that has recurred or is metastatic. This may include either single-agent or combination cytotoxic chemotherapy with radiotherapy or anti-EGFR treatment (eg, cetuximab). Adjuvant or neoadjuvant systemic chemotherapy does not count as a regimen for recurrent or metastatic disease.
* The subject has progressed within 6 months after completion of curative intent (definitive) treatment for localized/locoregionally advanced disease.
* The subject has not recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 Grade =1 from adverse events (AEs) due to investigational drugs or other medications that were administered more than 30 days before study enrollment with the sole exception of persistent Grade 2 peripheral neuropathy in patients who have previously received platinum-based therapy.
* The subject has known brain metastases.
* The subject has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active alcoholism, or psychiatric illness that would limit compliance with study requirements.
* The subject is pregnant or breastfeeding.
* The subject is known to be positive for the human immunodeficiency virus (HIV).
* The subject has an allergy or hypersensitivity to components of the GSK1363089 formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-08-27 (Actual); Primary Completion 2009-05-02 (Actual); Study Completion 2009-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (11):
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: MET111646 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MET111646 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MET111646 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MET111646 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: MET111646 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: MET111646 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MET111646 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 14 participants with advanced solid tumors were enrolled in this study. This study was conducted at up to 15 clinical sites in the United States.
Groups:
- Foretinib 240 mg: In each treatment period, participants received foretinib 240 milligram (mg) capsules orally on Days 1-5 of every 14-day cycle. Participants fasted 2 hours before to 1 hour after each dose. Each treatment cycle was 2 weeks. The 8-week study treatment period consisted of four 2-week treatment cycles. In the absence of progressive disease (PD) and unacceptable toxicity, participants may have received foretinib treatment on the same dosing schedule for up to 1 year at the discretion of the investigator, and beyond 1 year with the approval of the sponsor while participating in this study. During the treatment extension period, participants continued to receive foretinib on Days 1 through 5 followed by a 9-day observation period.
Period: Overall Study
Arm/Group | Foretinib 240 mg
Started | 14
Completed | 0
Not Completed | 14
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Not completed — Progressive Disease | 7
Not completed — Lost to Follow-up | 1
Not completed — Death | 1
Not completed — Participant non compliant with protocol | 1
Not completed — Decline in performance status | 1

BASELINE CHARACTERISTICS:
Groups:
- Foretinib 240 mg: In each treatment period, participants received foretinib 240 mg capsules orally on Days 1-5 of every 14-day cycle. Participants fasted 2 hours before to 1 hour after each dose. Each treatment cycle was 2 weeks. The 8-week study treatment period consisted of four 2-week treatment cycles. In the absence of PD and unacceptable toxicity, participants may have received foretinib treatment on the same dosing schedule for up to 1 year at the discretion of the investigator, and beyond 1 year with the approval of the sponsor while participating in this study. During the treatment extension period, participants continued to receive foretinib on Days 1 through 5 followed by a 9-day observation period.
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (8.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 13
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1
  White | 12
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Best Overall Response
Description: Best overall response was assessed by the investigator per response evaluation criteria in solid tumors (RECIST). Per RECIST v1.0 for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Tumor size was recorded at Baseline, and tumor response were recorded approximately every 8 weeks. Tumor response were classified by the investigator using RECIST criteria participant's best response whether observed in the study treatment period or the treatment extension period was considered. The best overall response was the best response recorded from the start of treatment until disease progression/recurrence. Number of participants who achieved best overall response were recorded.
Time Frame: Approximately up to 1 year
Population: safety population comprised of all participants who passed the screening criteria, enrolled in the study, and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 14
Participants
  Stable Disease | 7
  Progressive Disease | 3
  Unable to evaluate | 1

2. Primary Outcome: Percentage of Participants With Objective Response Rate (ORR)
Description: ORR was defined as the proportion of participants achieving best overall response of confirmed CR or PR divided by the total number of participants who received treatment. Per RECIST v1.0 for target lesions and assessed by MRI: CR, Disappearance of all target lesions; Partial Response PR, >=30% decrease in the sum of the longest diameter of target lesions; OR = CR + PR. Participants were evaluated for tumor response per RECIST. Percentage of participants with ORR were reported.
Time Frame: Approximately up to 1 year
Population: Safety Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 14
Percentage of participants | 0 [0 to 23.2]

3. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Data for number of participants who presented one or more adverse events (serious or non serious) was reported. An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Time Frame: Up to 20 months
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 14
Participants
  AEs, Any event | 14
  SAEs, Any event | 12

4. Primary Outcome: Number of Participants With Abnormalities of Common Toxicity Criteria for Adverse Events (CTCAE) Grade 3 in Laboratory Parameters (Clinical Chemistry and Hematology)
Description: The National Cancer Institute -CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each toxicity based on the following general guideline: Grade 1: Mild AE, Grade 2: Moderate AE, Grade 3: Severe AE, Grade 4: Life-threatening or disabling AE and Grade 5: Death related to AE. Number of participants with abnormalities of CTCAE grade 3 in clinical chemistry parameters: alanine aminotransferase (ALT), γ-glutamyl transferase (GGT), phosphate, low sodium and hematology parameters: Leukocyte and Lymphocytes were presented.
Time Frame: Up to 20 months
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 14
Participants
  Hematology, Leukocyte | 1
  Hematology, Lymphocytes | 2
  Serum chemistry, ALT | 1
  Serum chemistry, GGT | 2
  Serum chemistry, phosphate | 4
  Serum chemistry, low sodium | 2

5. Primary Outcome: Number of Participants With Abnormalities in Urinalysis
Description: Urinalysis parameters like appearance, color, pH, specific gravity, ketones, protein, glucose, bilirubin, nitrite, urobilinogen, and occult blood were performed. Number of participants with abnormalities are reported. In case of no abnormalities observed then it is reported as zero.
Time Frame: Week 5 [Day 29]
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 14
Participants | 0

6. Secondary Outcome: Duration of Progression-free Survival
Description: Progression-free survival was defined as the duration from the date of first dose to the date of disease progression or date of death without documented progression or date of study termination + 1. The start of confounding anticancer therapy was not treated as a censoring event. Time to progression or death was censored at the study termination date or at the analysis cutoff date, if earlier.
Time Frame: Approximately up to 1 year
Population: Safety Population.
Measure: Median (Full Range); unit: Months
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 14
Months | 3.65 [0.03 to 13.86]

7. Secondary Outcome: Duration of Overall Survival
Description: Overall survival was defined as the duration from the date of the first dose to the date of death. The start of a confounding anticancer therapy was treated as a censoring event. Every effort made to follow participant's until death. Time to death was censored at the date of the latest participant contact or at the analysis cutoff date, if earlier. Kaplan-Meier method was used to estimate the overall survival distribution.
Time Frame: Approximately up to 1 year
Population: Safety Population.
Measure: Median (Full Range); unit: Months
Groups:
- Foretinib 240 mg: This study consisted of a pre-treatment Period (screening and baseline evaluations), 8 week study treatment period, an optional treatment extension period, and a post-treatment period (including an end-of-treatment visit and an extended follow-up period). In each treatment period, participants received foretinib 240 mg capsules orally on Days 1-5 of every 14-day cycle. Participants fasted 2 hours before to 1 hour after each dose. Each treatment cycle was 2 weeks. The 8-week study treatment period consisted of four 2-week treatment cycles. In the absence of PD and unacceptable toxicity, participants may have received foretinib treatment on the same dosing schedule for up to 1 year at the discretion of the investigator, and beyond 1 year with the approval of the sponsor while participating in this study. During the treatment extension period, participants continued to receive foretinib on Days 1 through 5 followed by a 9-day observation period.
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 14
Months | 5.59 [2.46 to 15.57]

8. Secondary Outcome: Duration of Stable Disease
Description: Per RECIST v1.0 for target lesions and assessed by MRI: CR, Disappearance of all target lesions; Partial Response PR, >=30% decrease in the sum of the longest diameter of target lesions; OR = CR + PR. Duration of stable disease was defined as the time between the date of first dose of study drug and the first occurrence of 1 of the events: Tumor progression per RECIST as assessed by the investigator, Termination of study drug because of disease progression, Death due to disease progression, Disease progression as documented on the participant follow-up status form, Initiation of subsequent anticancer therapy.
Time Frame: Approximately up to 1 year
Population: Safety Population. Analysis set included only participants whose best overall response was not disease progression.
Measure: Median (Full Range); unit: Months
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 7
Months | 4.11 [1.81 to 13.86]

9. Secondary Outcome: Percentage Participants With Disease Stabilization Rate
Description: Disease stabilization rate was defined as the proportion of participants for whom the best overall response was a PR, CR, or stable disease. percentage participants with disease stabilization rate were presented.
Time Frame: Approximately up to 1 year
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 14
percentage of participants | 50.0 [23.0 to 77.0]

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Foretinib in Participants With Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Description: Plasma samples for pharmacokinetic analysis were planned to be drawn at time points: Day 1, 5, 19, 33, 43, 47 (approximately 15 minutes before dosing, and at 4 hours (±30 minutes) after dosing) of each treatment cycle, however these analyses were not completed. Cmax was defined as maximal measured plasma concentration over the time span specified. Data was not collected for this endpoint.
Time Frame: Day 1, 5, 19, 33, 43, 47 (pre-dose15 min) and 4 h (± 30 min) post-dose
Population: Safety population. Data was not collected for this endpoint.
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 0

11. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Foretinib in Participants With SCCHN
Description: tmax was defined as the time to the maximum or "peak" concentration of a drug observed after multiple administration. Blood samples were planned to be obtained during the time points: Day 1, 5, 19, 33, 43, 47 (approximately 15 minutes before dosing, and at 4 hours (±30 minutes) after dosing). However these analyses were not completed. Data was not collected for this endpoint.
Time Frame: Day 1, 5, 19, 33, 43, 47 (pre-dose15 min) and 4 h (± 30 min) post-dose
Population: Safety population. Data was not collected for this endpoint.
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 0

12. Secondary Outcome: Area Under the Concentration-time Curve (AUC) of Foretinib in Participants With SCCHN
Description: AUC was defined as area under the plasma concentration vs. time curve. Blood samples were planned to be collected on time points: Day 1, 5, 19, 33, 43, 47 (approximately 15 minutes before dosing, and at 4 hours (±30 minutes) after dosing). However these analyses were not completed. Data was not collected for this endpoint.
Time Frame: Day 1, 5, 19, 33, 43, 47 (pre-dose15 min) and 4 h (± 30 min) post-dose
Population: Safety population. Data was not collected for this endpoint.
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 0

13. Secondary Outcome: Elimination Half-life (t1/2) of Foretinib in Participants With SCCHN
Description: t1/2 was defined as the time to when half of the total amount of a particular substance is eliminated from the body. Blood samples were planned to be obtained during indicated time points: Day 1, 5, 19, 33, 43, 47 (approximately 15 minutes before dosing, and at 4 hours (±30 minutes) after dosing). However these analyses were not completed. Data was not collected for this endpoint.
Time Frame: Day 1, 5, 19, 33, 43, 47 (pre-dose15 min) and 4 h (± 30 min) post-dose
Population: Safety population. Data was not collected for this endpoint.
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 0

14. Secondary Outcome: Apparent Oral Clearance
Description: Blood samples were planned to be obtained during indicated time points: Day 1, 5, 19, 33, 43, 47 (approximately 15 minutes before dosing, and at 4 hours (±30 minutes) after dosing). Data for apparent oral clearance was not derived as pharmacokinetic analysis was not completed. Data was not collected for this endpoint.
Time Frame: Day 1, 5, 19, 33, 43, 47 (pre-dose15 min) and 4 h (± 30 min) post-dose
Population: Safety population. Data was not collected for this endpoint.
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 0

15. Secondary Outcome: Apparent Volume of Distribution
Description: Blood samples were planned to be obtained during indicated time points: Day 1, 5, 19, 33, 43, 47 (approximately 15 minutes before dosing, and at 4 hours (±30 minutes) after dosing). Data for apparent volume of distribution was not derived as pharmacokinetic analysis was not completed. Data was not collected for PK analysis.
Time Frame: Day 1, 5, 19, 33, 43, 47 (pre-dose15 min) and 4 h (± 30 min) post-dose
Population: Safety population. Data was not collected for this endpoint.
Arm/Group | Foretinib 240 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 20 months
Description: Safety Population was used to collect AE and SAE
Arm/Group | Foretinib 240 mg
All-Cause Mortality (participants affected / at risk) | 7/14
Serious Adverse Events (participants affected / at risk) | 12/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Foretinib 240 mg (N=14)
Dysphagia (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Foretinib 240 mg (N=14)
Constipation (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Stomach discomfort (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Swollen tongue (Gastrointestinal disorders) | 1
Tongue disorder (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 7
Mucosal inflammation (General disorders) | 4
Pain (General disorders) | 2
Pyrexia (General disorders) | 2
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Facial pain (General disorders) | 1
Local swelling (General disorders) | 1
Temperature intolerance (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Weight decreased (Investigations) | 4
Blood lactate dehydrogenase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood calcium decreased (Investigations) | 1
Heart rate increased (Investigations) | 1
Heart sounds abnormal (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Prothrombin time prolonged (Investigations) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 2
Amnesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Candidiasis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Panic attack (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 1
Wound secretion (Injury, poisoning and procedural complications) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Tachycardia (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.